CLINICAL TRIAL: NCT06708572
Title: Evaluation of the Use of Granulocyte Colony Stimulating Factor (GCSF) in Post Kasai Type 3 Biliary Atresia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCSFin biliary atresia
Record Dates: First submitted 2024-10-14; First posted 2024-11-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Granulocyte Colony-stimulating Factor; Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Protocol of cohort study will be conducted on 40 infants with the final diagnosis of biliary atresia type 3 (supported by the liver histology and intra-operative findings) divided into two groups one of them is for GCSF after Kasai operation, and the other group will be without GCSF therapy and their data will be collected retrospectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- biliary atresia without GCSF (No Intervention): 20 infants with the final diagnosis of biliary atresia type 3 (supported by the liver histology and intra-operative finding) for GCSF after Kasai operation will not receive GCSF.
- biliary atresia with GCSF (Experimental): 20 infants with the final diagnosis of biliary atresia type 3 (supported by the liver histology and intra-operative finding) for GCSF after Kasai operation will receive GCSF.
  Interventions: Drug: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Granulocyte Colony-Stimulating Factor — 20 patients will receive subcutaneous GCSF at a daily dose of 10ug/kg for 3 consecutive days. It is administered within 3-4 days after the Kasai procedure.
  Arms: biliary atresia with GCSF

SUMMARY:
The aim of the study is to evaluate the use of Granulocyte Colony Stimulating Factor (GCSF) on the clinical and biochemical outcome of type 3 biliary atresia post kasai.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a devastating disease manifest early in infancy characterized by bile duct injury and extrahepatic biliary obstruction, leading to cirrhosis in the majority of infants.

Although BA is a rare disease, occurring in ~1 in 5600 to 1 in 18,000 infants worldwide, it is considered the most common indication for liver transplantation in children.

However, despite a 50-60% rate of initial jaundice clearance, liver transplantation by 2 years of age is necessary for long term survival in many of the post-Kasai patients.

GCSF cytokine that stimulates neutrophil and hematopoietic stem cell (HSC) production and mobilization from the bone marrow, and has served as a complementary agent to bone marrow stem cell therapy for patients with congenital or acquired diseases of bone marrow suppression.

Granulocyte colony-stimulating factor (G-CSF) mobilizes CD34+(cluster of differentiation34) cells, these CD34+ cells increase hepatocyte growth factor inducing the proliferation of hepatic progenitor cells within 7 days.

In experimental liver diseases of toxin-induced or bile duct ligation-induced liver injury, GCSF-based stem cell therapy has the same effects as direct HSC transplantation on improving liver regeneration and suppressing the inflammatory and fibrotic responses to hepatic injury. The cellular and molecular mechanisms are unknown but are postulated to be derived from the many paracrine actions of GCSF.

ELIGIBILITY:
Inclusion Criteria:

* Infants with initial diagnosis of biliary atresia with biliary atresia score > 23.927 will be allocated for Kasai porto-enterostomy with intra-operative cholangiogram reaching type 3 biliary atresia anatomy as a final diagnosis.

Exclusion Criteria:

* Major cardiac, renal, pulmonary, neurological malformations or illnesses.
* Hemoglobinopathies, such as sickle cell anemia
* Active systemic infection.
* White blood cell count > 20,000 cells/mm3.
* Platelet count < 40,000 cells/mm3 or ≥ 800,000 cells/mm3.
* Purpura fulminans or unexplained vascular thrombotic conditions.

Ages: 20 Days to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with serum TBi (total bilirubin) ≥ 2 mg/dL at 3 months. | baseline
  Proportion of subjects with serum TBi (total bilirubin) ≥ 2 mg/dL at 3 months will be analyzed using generalized linear mixed effects model (GLMM) with a logistic link function for the covariates as fixed effects, with study sites as random effect to control for site variability in management practices and patient characteristics. The covariates are potential confounders for poor outcome, such as age at the time of Kasai, presence of ductal plate malformation, cholangitis and possibly CMV IgM(cytomegalovirus immune globulin M antibodies) positivity.

SECONDARY OUTCOMES:
Differences in the proportion of subjects with cholangitis at 6 months. | base line
  Differences in the proportion of subjects with cholangitis at 6 months will be calculated using the generalized linear mixed effect model with logistic link function for the covariates described in the primary outcome, with study sites as random effect to control for site variability in management practices and patient characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Cairo, Menofia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezerra JA, Wells RG, Mack CL, Karpen SJ, Hoofnagle JH, Doo E, Sokol RJ. Biliary Atresia: Clinical and Research Challenges for the Twenty-First Century. Hepatology. 2018 Sep;68(3):1163-1173. doi: 10.1002/hep.29905. PMID 29604222
- [Background] Overi D, Carpino G, Cardinale V, Franchitto A, Safarikia S, Onori P, Alvaro D, Gaudio E. Contribution of Resident Stem Cells to Liver and Biliary Tree Regeneration in Human Diseases. Int J Mol Sci. 2018 Sep 25;19(10):2917. doi: 10.3390/ijms19102917. PMID 30257529
- [Background] Corrado MM, Mack CL. Diagnostic Tools for Early Detection of Biliary Atresia: Is a Newborn Screen Attainable? Clin Liver Dis (Hoboken). 2022 Jan 24;19(1):25-28. doi: 10.1002/cld.1165. eCollection 2022 Jan. PMID 35106146